CLINICAL TRIAL: NCT05400785
Title: Efficacy of the Mobile Phone Application (Circadian Rhythms for Mood) for Prediction and Prevention of Mood Episode Recurrence in Mood Disorders Based on Machine Learning of Daily Digital Phenotype Variables : A Sham-controlled Randomized Clinical Trial
Brief Title: Efficacy of the Mobile Application for Prediction and Prevention of Mood Episode Recurrence Based on Machine Learning
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hucircadian (Industry)
Collaborators: Korea University Guro Hospital (Other); Korea University Ansan Hospital (Other); Pusan National University Hospital (Other); Inje University Ilsan Paik Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HC-CRM-01
Record Dates: First submitted 2022-05-27; First posted 2022-06-02 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Major Depressive Disorder; Bipolar 1 Disorder; Bipolar II Disorder
MeSH Terms: conditions — Depressive Disorder, Major; Bipolar Disorder | interventions — Circadian Rhythm; picolinic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Active CRM (Active Comparator)
  Interventions: Other: Circadian Rhythms for Mood (CRM) application - Active
- Sham CRM (Sham Comparator)
  Interventions: Other: Circadian Rhythms for Mood (CRM) application - Sham

INTERVENTIONS:
Other: Circadian Rhythms for Mood (CRM) application - Active — The study subjects participating in this clinical trial wear wearable activity tracker 24 hours a day for a continuous period of time and run the CRM app once a day to check their conditions (feelings, vitality, sleep, etc.) in the Daily Symptom Assessment (eMoodChart). The active intervention group are provided with mood prediction results and instructions as feedback through the 'life report' and push notification in the application.
  Arms: Active CRM
Other: Circadian Rhythms for Mood (CRM) application - Sham — The study subjects assigned to the sham intervention group are provided with feedbacks operated by dummy algorithm. The application is visually indistinguishable from active CRM, and it is designed to minimize behavioral change.
  Arms: Sham CRM

SUMMARY:
This study was designed to evaluate the efficacy of the mobile application named Circadian Rhythm for Mood (CRM), which was developed to prevent recurring episodes of mood disorders (major depressive disorders, bipolar disorders type 1 and 2) based on machine learning.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, 19-70 years old
* Diagnosis with Bipolar I disorder, Bipolar II disorder, Major depressive disorder based on DSM-5 criteria, in euthymic state for more than two weeks at the time of the recruitment
* Android smartphone users, capable of installing and executing the CRM application
* Consent to wear wearable device (Fitbit) continuously and synchronize and backup data regularly

Exclusion Criteria:

* Patients who have not experienced major depressive, manic, or hypomanic episode in the last two years
* Patients who are difficult to specify mood episode or evaluate symptoms of mood episode independently due to personality traits (borderline personality trait, cyclothymic temperament, etc.)
* Patients with degenerative neurological disorders (Parkinson's disease, dementia, Huntington's disease, etc.), neurodevelopmental disorders (intellectual disorder, autism spectrum disorder, down syndrome, etc.), epilepsy, severe traumatic brain damage, stroke, and other brain neurological disorders
* Inmates or patients who are forced into custody for the treatment of mental or physical illness (non-voluntary isolation or hospitalization)
* Patients with difficulties in understanding the objectives and process of the study and the potential benefits and risks of participating in the study

Ages: 19 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 93 (Actual)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-12-21 (Actual); Study Completion 2023-12-21 (Actual)

PRIMARY OUTCOMES:
Comparison of total number of recurrent mood episodes between the active and sham groups | 12 months
  We aim to evaluate the efficacy of reducing recurrence rate of mood episodes through the CRM mobile application.
Comparison of duration of mood episodes between the active and sham groups | 12 months
  We aim to evaluate the efficacy of reducing duration of mood episodes through the CRM mobile application.

CONTACTS AND LOCATIONS:
Locations (1):
- Korea University Anam Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Yeom JW, Yoon Y, Seo JY, Cho CH, Lee T, Lee JB, Jeon S, Kim L, Lee HJ. Daily Self-Monitoring and Feedback of Circadian Rhythm Measures in Major Depression and Bipolar Disorder Using Wearable Devices and Smartphones-The Circadian Rhythm for Mood (CRM(R)) Trial Protocol: A Randomized Sham Controlled Double-Blind Trial. Psychiatry Investig. 2024 Aug;21(8):918-924. doi: 10.30773/pi.2024.0133. Epub 2024 Aug 2. PMID 39086163